CLINICAL TRIAL: NCT04488445
Title: Acute Effects of Strength Training Over Executive Functions in Adolescents: A Randomized Controlled Trial
Brief Title: Strength Training and Executive Functions: A Randomized Controlled Trial
Acronym: ASTOEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Rubén López-Bueno, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UZaragoza13091978
Record Dates: First submitted 2020-07-18; First posted 2020-07-28 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Executive Function Disorder; Strength Training; Adolescent Behavior; Academic Achievement
MeSH Terms: conditions — Adolescent Behavior | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training (Experimental): The intervention group performs a resistance training based on a resistance exercise of 3 sets of 3 to 5 repetitions (90% of an estimated 1 RM) and 3 minutes of resting time between sets.
  Interventions: Behavioral: Strength training
- Stretching (Placebo Comparator): The control group performs 3 exercises of stretching and balance during one minute each and three sets. One minute of resting time between sets.
  Interventions: Behavioral: Stretch and balance training

INTERVENTIONS:
Behavioral: Strength training — 3 sets of 3 to 5 repetitions with 4 minutes of rest between sets. 90% load of 1 maximum repetition of a resistance exercise
  Other Names: Resistance training
  Arms: Strength Training
Behavioral: Stretch and balance training — 3 sets of 3 exercises of stretching and balance of one minute each. One minute of resting time between sets.
  Other Names: Stretching
  Arms: Stretching

SUMMARY:
A group of 50 age-schooled adolescents was randomized into one intervention and another control group of 25 subjects each. After estimating one maximum repetition for all the participants in a previous session, the intervention group performed a resistance training based on a resistance exercise of 3 sets of 3 to 5 repetitions (90% of an estimated 1 RM) whereas the control group performed both stretching and balance exercises. Measures of executive functions ( i.e. a cognitive function associated with academic performance) were taken for all the participants before and after the training. Both independent and paired t-test will serve to check differences between and within groups respectively.

DETAILED DESCRIPTION:
A group of 50 age-schooled adolescents was randomized into one intervention and another control group of 25 subjects each. After estimating one maximum repetition for all the participants in a previous session, the intervention group performed a resistance training based on a resistance exercise of 3 sets of 3 to 5 repetitions (90% of an estimated 1 RM) whereas the control group performed both stretching and balance exercises. Measures of executive functions ( i.e. a cognitive function associated with academic performance) were taken for all the participants before and after the training. Both independent and paired t-test will serve to check differences between and within groups respectively. The selected resistance exercise is based on a global muscle involvement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy age-schooled adolescent

Exclusion Criteria:

* Not healthy, injured age-schooled adolescent

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Time to successfully complete the executive function test | up to 24 weeks
  Executive function

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Calatayud, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Zaragoza, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No